CLINICAL TRIAL: NCT07132658
Title: PROJECT#2: MRI-guided Local SBRT Prostate Program
Brief Title: MRI-guided Ultrahypofractionated SBRT Prostate Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2024.198
Record Dates: First submitted 2025-06-19; First posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; NCCN Low Risk; NCCN Favorable Intermediate Risk
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Initial Phase (Active Comparator): Whole Gland 36.25Gy/5Rx
  Interventions: Radiation: MR-Guided SBRT
- Study Phase (Experimental): Whole Gland 27Gy/2Rx
  Interventions: Radiation: MR-Guided SBRT
- Final Phase (Experimental): Asymmetrical Whole Gland 27Gy/2Rx
  Interventions: Radiation: MR-Guided SBRT

INTERVENTIONS:
Radiation: MR-Guided SBRT — MR-Guided SBRT

SUMMARY:
The goal of this clinical trial is to learn if the use of MRI-guided asymmetric ultrahipofractionated irradiation (2 fractions with dose increase in the tumor areas and dose sparing in urethra, rectum and neurovascular bundles) produces similar results in terms of local control and complications to standard 5-fraction SBRT.

DETAILED DESCRIPTION:
The implementation of Magnetic Resonance Image Guided Radiotherapy (MRgRT) into a Prostate Cancer Program aims to reproduce the results obtained with state-of-the-art brachytherapy or EBRT with the added advantage of convenience and lack of invasiveness.

ELIGIBILITY:
Optimal Inclusion Criteria

* Patients with low to favorable intermediate-risk prostate cancer as per the NCCN stratification criteria .
* No prior radiation therapy to the target areas
* Expected patient survival >5 years
* Patient able to undergo a MRI exam

Cautionary Inclusion Criteria

* Suboptimal candidates for high-dose therapy such as elderly, frail patients or patients with large volume glands (i.e, >60cm3) or extensive TURP in the prior 6-12 months should be considered cautionary indications.
* Patients with higher risk but low volume disease not candidates for ENI may be treated on an individual basis

Exclusion Criteria

* Prior radiation therapy to the target areas
* Expected patient survival below 5 years
* Patient unable to undergo a MRI exam

Ages: 18 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2030-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Biochemical Relapse-Free Survival | 5-years
  To achieve a 4-year biochemical relapse-free survival of 95%.
Adverse Events | 5-years
  To decrease urinary grade 3 or greater toxicity below 3% and rectal grade 3 or greater toxicity below 1%.

SECONDARY OUTCOMES:
Quality of Life (QOL) assessment | 5-years
  Determination of QOL with International Prostate Symptom Score (IPSS) and European Organisation for Research and Treatment of Cancer (EORTC) quality of life questionnaire (QLQ)-PR25. IPSS ranges from 0 to 35 with higher values representing worse functioning. EORTC QLQ PR-25 ranges from 0-100 with higher values representing better functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Martínez-Monge, M.D., Principal Investigator — Clínica Universidad de Navarra; Luis Fuertes, M.D., Principal Investigator — Clínica Universidad de Navarra

IPD SHARING:
Plan to Share IPD: Yes
On request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Jul 1st, 2025 to June 30, 2030
Access Criteria: On request